CLINICAL TRIAL: NCT03196570
Title: Increasing Physical Activity in Latino Men Through Tailoring
Brief Title: Increasing Physical Activity in Latino Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Kim Gans, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1612001664
Record Dates: First submitted 2017-06-15; First posted 2017-06-23 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After randomization into the intervention arm, participants will be instructed on how to use the Spanish language study website. During the six month intervention, they will complete online questionnaires to determine their stage of change towards increasing physical activity. A manual of information will be automatically generated based on their responses. Participants can read this information online, along with tip sheets related to increasing physical activity. On the website they can also set weekly goals and log their weekly PA. It will also include short videos with demonstrations for PA they can do at home and around their neighborhood. Information will also include community resources (community centers, public events, parks) where they can be physically active. Participants will also receive prompts and encouragement via text-message to encourage them to log into the website and continue to track their progress.
  Interventions: Behavioral: Physical Activity Intervention
- Contact Control (Active Comparator): Participants in the control arm will attend the same baseline orientation sessions and measurements as the intervention arm. After randomization into the control group, participants will complete an introductory in-person session to introduce them to a website, similar in design, with information on health topics other than physical activity, including diet and other factors associated with CVD risk. It will include information from NHLBI heart health materials for Latinos. Topics include healthy eating, increasing fruit and vegetable consumption, reducing fat and salt intake, learning about cholesterol, stress management. Participants will log onto a separate website unique to the control group and complete monthly surveys on the wellness topics and their progress. Participants will also receive prompts and encouragement text-messages to encourage them to log onto the website.
  Interventions: Behavioral: Wellness Contact Control

INTERVENTIONS:
Behavioral: Physical Activity Intervention — After randomization into the intervention arm, participants will be instructed on how to use the Spanish language study website. During the six month intervention, they will complete online questionnaires to determine their stage of change towards increasing physical activity. A manual of information will be automatically generated based on their responses. Participants can read this information online, along with tip sheets related to increasing physical activity. On the website they can also set weekly goals and log their weekly PA. It will also include short videos with demonstrations for PA they can do at home and around their neighborhood. Information will also include community resources (community centers, public events, parks) where they can be physically active. Participants will also receive prompts and encouragement via text-message to encourage them to log into the website and continue to track their progress.
  Arms: Intervention
Behavioral: Wellness Contact Control — Participants in the control arm will attend the same baseline orientation sessions and measurements as the intervention arm. After randomization into the control group, participants will complete an introductory in-person session to introduce them to a website, similar in design, with information on health topics other than physical activity, including diet and other factors associated with CVD risk. It will include information from NHLBI heart health materials for Latinos. Topics include healthy eating, increasing fruit and vegetable consumption, reducing fat and salt intake, learning about cholesterol, stress management. Participants will log onto a separate website unique to the control group and complete monthly surveys on the wellness topics and their progress. Participants will also receive prompts and encouragement text-messages to encourage them to log onto the website.
  Arms: Contact Control

SUMMARY:
The purpose of this study is to determine the feasibility and preliminary efficacy of a web and text-messaged based intervention designed to increase physical activity among Latino men in Rhode Island. The study will also examine potential moderators of treatment effects including demographics, acculturation, and environmental variables such as the neighborhood built, social and economic environments.

DETAILED DESCRIPTION:
Physical Activity in Latino Men Through Tailoring is an individually randomized web and text message based pilot study, designed to increase physical activity amongst Latino men. The study is conducting formative research with a diverse population of Latino men to inform the adaptation of the Pasos Hacia La Salud web-based intervention, which was developed for Latina women, to an intervention focused on Latino men. Consideration will also be taken to ensure intervention material is culturally appropriate for Latino men of Caribbean, South and Central American origin. Half the study participants will be randomized into the intervention arm and half into the comparison group. Participants in the intervention arm will have access to a website where they can complete questionnaires, receive information, log their physical activity and set goals. Participants complete monthly questionnaires to establish their stage of change toward increasing their physical activity and receive information manuals based on their current stage of change. They will also have access to tip sheets via the study website and receive reoccurring text messages reminding them to log into the website. Participants in the comparison arm will have access to a similar website with information related to nutrition and overall wellness, not including physical activity.

The primary aims of this project are (1) to conduct formative research with a diverse population of RI Latino men to adapt the existing web-based interventions and add text message-based components to complement and enhance the intervention. The second primary aim is to determine the feasibility, acceptability, and preliminary efficacy of the intervention and the study recruitment, implementation and evaluation protocols with a diverse population of Latino men. An additional exploratory aim will be to examine potential moderators of treatment effects including demographics, acculturation, and environmental variables such as the neighborhood built, social and economic environments. The hypothesis is that participants randomized to the intervention condition will have greater increases in weekly minutes of physical activity after six months than those randomized to a wellness control condition. The results of this pilot study will inform a future randomized controlled trial with Latino men to increase PA.

ELIGIBILITY:
Inclusion Criteria:

* Be sedentary ( participate in moderate intensity leisure time PA two days a week for less than 30 minutes a day, or less)
* Identify as a Latino male
* Speak Spanish
* Score of more than 16% on Spanish Shortened Test of Functional Health Literacy in Adults
* Own a cell phone with texting capabilities and have internet access

Exclusion Criteria:

* History of myocardial infarction or angina, insulin-dependent diabetes or hospitalization for diabetes in the past year, stroke, osteoarthritis, osteoporosis, orthopedic problems, or any medical condition that would make PA unsafe.
* Planning to move from the area in the next 6 months
* Hospitalization due to a psychiatric disorder in the past 3 years.
* BMI of 45 or higher and/or taking any medication that may impair PA tolerance or performance.
* If they or another family member is already enrolled in another PA or weight control study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity from Baseline to 6 months | Baseline and 6 months
  Minutes of Moderate and Vigorous Physical Activity

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dulin AJ, Dunsiger S, Benitez T, Larsen B, Marcus BH, Champion G, Gans KM. The Hombres Saludables Physical Activity Web-Based and Mobile Phone Intervention: Pilot Randomized Controlled Trial With Latino Men. J Med Internet Res. 2023 Dec 7;25:e39310. doi: 10.2196/39310. PMID 38060285
- [Derived] Gans KM, Dulin A, Palomo V, Benitez T, Dunsiger S, Dionne L, Champion G, Edgar R, Marcus B. A Tailored Web- and Text-Based Intervention to Increase Physical Activity for Latino Men: Protocol for a Randomized Controlled Feasibility Trial. JMIR Res Protoc. 2021 Jan 29;10(1):e23690. doi: 10.2196/23690. PMID 33512327